CLINICAL TRIAL: NCT01336517
Title: Comprehensive Evaluations of the Effect of an Ankle Foot Orthoses for Ambulatory Function in Adults With Hemiplegia
Brief Title: Evaluation of the Effect of an Ankle Foot Orthoses for Ambulatory Function
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Karen Nolan, Ph.D., Kessler Foundation Research Center
Other Study IDs: E59007
Record Dates: First submitted 2009-10-02; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Hemiplegia, Spastic
Keywords: Stroke; Hemiplegia; AFO; Gait
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this investigation is to evaluate the effect of a lower leg brace on walking efficiency and community walking in people who have weakness in one side of the body caused after a stroke. The evaluation will consist of several tests that will evaluate movement, tightness, balance and sensation in affected leg.

DETAILED DESCRIPTION:
To comprehensively evaluate the effect of an AFO on ambulatory function and loading in hemiplegic gait. This study is addressing important questions regarding the effect of an AFO on gait and introduces technology for quantifiable objective assessment of AFO effectiveness. It will attempt to identify if AFO wear compliance increases community ambulation and walking efficiency bilaterally. Research is needed to fully understand how compliance affects mobility outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75
* Have sustained a stroke at least 6 months prior to study enrollment
* Use a prescribed custom brace while walking
* Have no history of injury, orthopedic or other medical problem in the normal leg
* Be able to walk independently or with close supervision for 25 feet without a brace or cane
* Wear shoes sizes 5 1/2 - 11 US womens or size 6-13 US mens

Exclusion Criteria:

* Orthopedic problems or history that will interfere with walking or limit the range of motion of legs
* Neurological illness, history, or conditions that my interfere with walking except for stroke
* Psychiatric conditions or history that would interfere with the ability to walk or follow directions
* Serious lung or heart condition that could severely limit the ability to walk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a history of hemiplegia secondary to stroke, between the ages of 18 and 75, who are greater than 6 months post and have been prescribed a custom molded AFO for assistance with gait deviations
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Nolan, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States